CLINICAL TRIAL: NCT03178409
Title: Survival After Hepatectomy for Combined Hepatocellular Cholagiocarcinoma
Brief Title: Combined HCC-MFCCC
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Director of the Department of Hepatobiliary and General Surgery, University of Milan
Other Study IDs: cHCC-MFCCC
Record Dates: First submitted 2017-06-04; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Liver Carcinoma; Hepatocellular Carcinoma; Cholangiocarcinoma; Surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cHCC-MFCCC: Patients affected by combined HCC-MFCCC
  Interventions: Procedure: Hepatectomy
- HCC: Patients affected by classical HCC
  Interventions: Procedure: Hepatectomy
- MFCCC: Patients affected by classical MFCCC
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy — Removal of a part of the liver
  Other Names: Liver resection; Liver surgery

SUMMARY:
Combined hepatocellular and mass-forming cholangiocarcinoma (cHCC-MFCCC) is a rare tumor. The aim of this study was the analysis of the outcome comparing such tumor with classic hepatocellular carcinoma (HCC) and mass-forming cholangiocarcinoma (MFCCC).

DETAILED DESCRIPTION:
The institutional prospectively maintained database was queried, and 20 patients with cHCC-MFCCC were identified. A 2:1 match was performed with 40 patients operated in the same period for HCC, and with 40 operated for MFCCC. Only T1 or T2 patients N0 M0 were considered. Primary endpoint was the overall survival (OS) and disease-free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

* positive histology for cHCC-MFCCC, HCC, and MFCCC
* complete clinical, surgical, pathological and follow-up data.

Exclusion Criteria:

* patients preoperatively treated with chemotherapy, radiofrequency ablation or trans-arterial therapies were excluded.
* patients operated for recurrent disease and/or with non-radical surgery
* patients with missing data were also excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by cHCC-MFCCC, or HCC or MFCCC.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Survival analysis | From 3 months after surgery up to 60 months after surgery
  Analysis of overall and disease-free survival of patients resected for cHCC-MFCCC versus those resected for HCC versus those resected for MFCCC

IPD SHARING:
Plan to Share IPD: No